CLINICAL TRIAL: NCT00422643
Title: The Effect of Intraaricular Knee Injections of Hyaluronic Acid (HA) on Bone and Cartilaginous Debris, as a Therapeutic Indicator
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Collaborators: Ferring Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: DEBICTIL
Record Dates: First submitted 2007-01-15; First posted 2007-01-17 (Estimated); Last update posted 2007-01-18 (Estimated); Status verified 2007-01

CONDITIONS: Osteoarthritis of the Knee
Keywords: OA,HA,Intra-articular
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Hyaluronic Acid

INTERVENTIONS:
Drug: Sodium hyaluronate (hyaluronic acid)

SUMMARY:
Osteoarthritis is the most common disease effecting human beings with incidence of about 20% and prevalence close to 80% of the adult population. It is most common after the age of 60 years and more in females with the ratio 4:1 F:M. Osteoarthritis Can be present in every hyaline joint, but is mostly damaging to the weight bearing joints, the knees and hips. At the final stage of cartilage destruction (from wear and tear) joint replacement is the solution. Since these operations were introduced about 50 years ago, the indications and the number of yearly procedures has been increasing with alarming speed. Last year in the united states, about 500,000 Total Knee procedures were done, exceeding Total Hip replacements.

By 2030, close to 4.5 million joint replacement procedures are expected in the United States, the majority of which will be knee replacements. Joint replacement is the solution for the final stage of damaged cartilage. In early and advanced stages of cartilage wear and specifically in the knee H.A. acts as an anti inflammatory and lubricant agent, reducing the knee pain and improving knee motion and function.

The biological effect of H.A. is well documented in clinical studies and less with scientific evidence derived from patients themselves.

Our study proposal briefly is, as follows:

60 patients with evidence of osteoarthritis of the knees will join the study after I.R.B. (Helsinki Committee) approval. All of them will be examined, x-rays will be performed and blood tests will exclude patients with infections or inflammatory disease. A V.A.S. (Visual Analog Score) and SF-36 evaluation form will be completed prior to each intraarticular injection, in addition to a complete medical examination. The enrolled patients will receive the usual three intraarticular knee injections of H.A.(Arthrease), but prior to each injection, the joint will be aspirated and the joint fluid will be analyzed for Chondroitin sulfate type I and type II as described further in this project.

Three and six months after the third initial injections, the patients will recalled and joint fluid will be aspirated again, followed by an H.A. injections, if symptomatic.

This study is the only one ever proposed, for evaluating joint debris qualitatively and quantitatively. It will provide clinical information as well as objective data on the preservation of the joint cartilage. Hopefully, this study will provide additional information such as the relationship between the presence of debris and symptomatic vs. asymptomatic patients. It may help in determining how long the injected H.A. has an effect and whether serial and periodical injections are indicated.

Inclusion criteria:

1. patients with the diagnosis of Osteoarhtritis of the knee, graded according to Kellgren as grade 1-4

Exclusion criteria:

1. Patients that suffer from acute septic arthritis.
2. Patients that treated with coumadin and/or other anti-coagulant drugs
3. Patients that show mental or physical conditions, which preclude compliance with study and/or device.

ELIGIBILITY:
Inclusion criteria:

* Patients with the diagnosis of Osteoarhtritis of the knee, graded according to Kellgren as grade 1-4

Exclusion criteria:

* Patients that suffer from acute septic arthritis.
* Patients that treated with coumadin and/or other anti-coagulant drugs
* Patients that show mental or physical conditions, which preclude compliance with study and/or device.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2007-03; Study Completion 2007-10

PRIMARY OUTCOMES:
To provide additional information such as the relationship between the presence of debris and symptomatic vs. asymptomatic patients.
Determining how long the injected H.A. has an effect and whether serial and periodical injections are indicated.

CONTACTS AND LOCATIONS:
Overall Officials: ronen debi, md, Principal Investigator — assaf harofe medical center
Locations (1):
- Orthopedic, Ẕerifin, Israel